CLINICAL TRIAL: NCT00471718
Title: A Phase1/2 Trial of ABT-751 in Patients With Advanced, Androgen-Independent Prostate Cancer
Brief Title: ABT-751 in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: pharmaceutical company closed study because the treatment was not effective
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey A. Sosman, MD, Professor of Medicine; Director, Melanoma and Tumor Immunotherapy, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC URO 0426; VU-VICC-URO-0426
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ABT751

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I/II: Chemotherapy ABT-751 (Experimental): Phase I: Patients receive oral ABT-751 twice daily on days 1-7 and 15-21.
  Phase II: Patients receive ABT-751 twice daily
  Interventions: Drug: ABT-751

INTERVENTIONS:
Drug: ABT-751 — Phase I:
  Cohort | Number of Patients |Dose (mg) ABT-751 (BID)
  * -1 | 3-6 |100 mg BID
  * 1 | 3-6 |125 mg BID
  * 2 | 3-6 |150 mg BID
  * 3 | 3-6 |175 mg BID
  * 4 | 3-6 |200 mg BID
  Phase II:
  Patients receive ABT-751 at 125mg po BID for 7 days on, 7 days off (X2) for a 28 day cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ABT-751, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ABT-751 and to see how well it works in treating patients with metastatic prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and efficacy of ABT-751 in patients with androgen-independent, hormone-refractory metastatic prostate cancer and determine the maximum tolerated dose (MTD) and optimal phase II dose of this drug in these patients.

Secondary

* Determine the objective response rate (partial and complete response) in patients with measurable disease treated with this drug.
* Evaluate the effect of this drug on prostate-specific antigen (PSA) response in patients with nonmeasurable disease.
* Determine the time to tumor progression in patients treated with this drug.
* Determine survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

* Phase I: Patients receive oral ABT-751 twice daily on days 1-7 and 15-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ABT-751 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 50 additional patients may be treated at the recommended phase II dose (RPTD) which is the dose level at the maximally administered dose.

* Phase II: Patients receive ABT-751 at the MTD determined in phase I. After completion of study treatment, patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Patients must have histologically proven adenocarcinoma of the prostate gland.
* Patients must have metastatic disease (e.g. bone metastases, pelvic mass, nodal, liver or lung metastases), with evidence of radiographic progression (including bone scans observed during last treatment) or serologically -Patients with bone-only metastases (i.e. lacking soft tissue or visceral disease) must have a PSA level > 10 ng/mls. Patients with soft tissue metastases and/or visceral disease must have either measurable disease OR a PSA level > 10 ng/ml.
* Patients must have had prior treatment with bilateral orchiectomy or other primary hormonal therapy (e.g. LHRH therapy, estrogens, etc.) with evidence of treatment failure and simultaneous documentation of a castrate testosterone level (< 50 ng/dL) NOTE: Patients who have not undergone bilateral orchiectomy must continue LHRH agonist therapy for the duration of this protocol unless this medically contraindicated.
* For patients previously treated with flutamide, nilutamide, or bicalutamide: patients must have discontinued flutamide or nilutamide > 4 weeks prior to randomization (> 6 weeks for bicalutamide) with no evidence of an anti-androgen withdrawal response (i.e. no decline in serum PSA and/or no improvement in baseline scans).
* Patients must have received prior therapy with docetaxel alone or in combination with either prednisone or estramustine. This therapy may have been given in a neoadjuvant, adjuvant or metastatic setting
* Patients must not have received radiotherapy < 3 weeks prior to randomization. If patients have received prior radiotherapy to an evaluable lesion(s), there must be evidence of radiographic progression prior to entry.
* Patients must not have received prior Strontium 89, Samarium 153, or other therapeutic radioisotopes.
* Patients must have recovered from all systemic toxicities due to prior treatment for prostate cancer (does not include incontinence, impotence, etc. secondary to primary therapy)
* The patient must have an ECOG Performance Status of 0-1
* The patient must have adequate hematologic, renal and hepatic function as follows:

  1. Hematologic: ANC > 1200/mm3; hemoglobin > 9.0 g/dl; platelets > 100,000/mm3
  2. Renal: serum creatinine < 2.0 mg/dL
  3. Hepatic: bilirubin < 2.5 mg/dL; AST and ALT < 2.5X upper limit of normal (ULN); < 5X ULN for patients with hepatic metastases
* Sexually-active patients must use a contraceptive method deemed acceptable by the investigator while in the study and for up to 3 months following completion of therapy.
* The patient or the patient's legally acceptable representative has voluntarily signed and dated an informed consent approved by and Institutional Review Board prior to any study any study specific procedures.
* Patients may be receiving bisphosphonate therapy prior to randomization and continue while receiving protocol therapy, but must not begin treatment with bispohosphonates while receiving protocol therapy. Patients on bisphosphonates must have completed at least 4 weeks of bisphosphonate therapy prior to entry onto study.
* Patients with a history of a prior malignancy are eligible provided they were treated with curative intent and have been free of disease for the time period considered appropriate for the specific malignancy.

Exclusion Criteria:

* No active angina pectoris, uncontrolled hypertension, or known heart disease of New York Heart Association Class III-IV. Patients must not have a history of myocardial infarction, congestive cardiac failure (New York Heart Association Class 3), or coronary angioplasty/stenting < 6 months prior to entry.
* No carcinomatous meningitis or brain metastases.
* Any investigational therapy within 4 weeks.
* No serious concurrent medical illness or active infection, which, in the opinion of the investigator, would jeopardize the ability of the patient to receive the chemotherapy outlined in this protocol with reasonable safety.
* Documented history of allergy to sulfa medications.
* Current colchicines treatment
* Greater than Grade 1 CTC neurology category findings (Appendix A).
* Prior treatment with more than 1 prior chemotherapy regimen.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Sosman, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study began enrolling October 2004 through December 2007.
Pre-assignment Details: A total of 34 patients were consented in Phase I and Phase II, 7 of which were not eligible.
Groups:
- Phase I/II: ABT-751: Phase I: Patients receive oral ABT-751 twice daily on days 1-7 and 15-21. Phase II: Patients receive ABT-751 at 125mg twice daily, 7 days on, 7 days off (x2)for a 28-day cycle
Period: Overall Study
Arm/Group | Phase I/II: ABT-751
Started | 27
Completed | 0
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — other complicating disease | 1
Not completed — disease progression | 22
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phase I/II: ABT-751
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is determined by the 3+3 study design, in which patients are enrolled in cohorts of 3. In any dose cohort, if 1 patient of 3 experience dose-limiting toxicity (DLT), three additional patients will be enrolled at the same dose level. Whenever >=2 of 6 subjects experience a DLT, then the maximum tolerated dose (MTD) has been exceeded. The MTD is generally one dose below that at which DLT occurs in >= 2 of 6 subjects in any given cohort.
Time Frame: up to four weeks
Population: Phase I patients who received treatment
Measure: Number; unit: mg twice a day
Groups:
- ABT-751: Phase I: Patients receive oral ABT-751 twice daily on days 1-7 and 15-21. Phase II: Patients receive ABT-751 at 125mg twice daily, 7 days on, 7 days off (x2)for a 28-day cycle
Arm/Group | ABT-751
Number analyzed (Participants) | 17
mg twice a day | 125

2. Secondary Outcome: Number of Patients With Objective Response (CR & PR) by RECIST
Description: Number of participants in each best tumor response category, RECIST criteria (v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in sum longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in sum LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of smallest sum of the LD of target lesions.
Time Frame: after four weeks
Population: Participants with measurable disease who completed at least one cycle of treatment with tumor assessment.
Measure: Number; unit: participants
Groups:
- Phase I/11: ABT-751: Duration of overall response from time measurements are met for CR or PR until date that recurrence or PD is objectively documented
Arm/Group | Phase I/11: ABT-751
Number analyzed (Participants) | 6
participants
  Complete Response | 0
  Partial Response | 0

3. Secondary Outcome: Median Time to Tumor Progression
Description: Number of weeks from the date the patient started study drug to the date of the patient's tumor progression documented radiographically or by PSA testing.
  Tumor progression is measured at baseline and after two 28-day cycles
Time Frame: date on study to date of progression
Population: Patients who received treatment and who were available for measurement of tumor or who available for PSA testing
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase I/II: ABT-751
Number analyzed (Participants) | 19
Weeks | 4 [3.83 to 4.17]

4. Secondary Outcome: Overall Survival
Description: Number of weeks from the date the patient started study drug to the date of the patient's death.
Time Frame: date on study to date of death from any cause
Population: At the time of this analysis, all 27 patients were deceased due to progressive prostate cancer.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase I/II: ABT-751
Number analyzed (Participants) | 19
Weeks | 35.3 [26.4 to 44.2]

5. Secondary Outcome: Safety Profile Based on Number of Patients With Worst Grade Toxicities
Description: Not all participants necessarily have an adverse event, thus not everyone will be accounted for in worst-grade toxicities. Likewise, one participant can potentially have more than one event in various grades 1-5 which accounts for the difference in number of patients analyzed and total number in the worst-grade toxicity tables. Tables represent the number of patients with worst-grade toxicity at each of five grades (grade 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening or disabling, grade 5 = death)following NCI Common Toxicity Criteria
Time Frame: at 30 days after final treatment dose
Measure: Number; unit: patients
Arm/Group | Phase I/II: ABT-751
Number analyzed (Participants) | 27
patients
  No. of patients with worst-grade toxicity of 1 | 0
  No. of patients with worst-grade toxicity of 2 | 10
  No. of patients with worst-grade toxicity of 3 | 14
  No. of patients with worst-grade toxicity of 4 | 3
  No. of patients with worst-grade toxicity of 5 | 0

6. Primary Outcome: Number of Patients Who Demonstrated Treatment Effectiveness Based on Prostate Specific Antigen (PSA) Response in Non-measurable Disease
Description: Patients with a minimum 50% decline in PSA from pre-treatment baseline, confirmed by a second PSA 4 or more weeks later, measured in nanograms per milliliter of blood.
Time Frame: after four weeks
Population: Men with non-measurable disease: all other lesions, bone lesions, leptomeningeal disease, cystic lesions, abdominal masses that are not followed by imaging techniques
Measure: Number; unit: participants
Groups:
- Phase I/11: ABT-751: Phase I: Patients receive oral ABT-751 twice daily on days 1-7 and 15-21. Phase II: Patients receive ABT-751 at 125mg twice daily, 7 days on, 7 days off (x2)for a 28-day cycle
Arm/Group | Phase I/11: ABT-751
Number analyzed (Participants) | 19
participants | 0

ADVERSE EVENTS:
Arm/Group | Phase I/II: ABT-751
Serious Adverse Events (participants affected / at risk) | 7/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II: ABT-751 (N=27)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pain, tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
hemoglobin (Blood and lymphatic system disorders) | 2 (2)
mood alteration (Psychiatric disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
hyperglycemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
confusion (Psychiatric disorders) | 2 (2)
neuropathy cranial (Nervous system disorders) | 1 (1)
neuropathy motor weakness (Nervous system disorders) | 1 (1)
speech impairment (Nervous system disorders) | 1 (1)
extrapyramidal (Nervous system disorders) | 1 (1)
fever (General disorders) | 1 (1)
Infection with normal ANC (Infections and infestations) | 1 (1)
memory impairment (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II: ABT-751 (N=27)
Constipation (General disorders) | 15 (26)
neuropathy (Nervous system disorders) | 13 (21)
pain (General disorders) | 18 (36)
anemia (Blood and lymphatic system disorders) | 18 (26)
hyperglycemia (Metabolism and nutrition disorders) | 15 (21)
gastrointestinal disorders (Gastrointestinal disorders) | 11 (16)
fatigue (General disorders) | 19 (35)
anorexia (Psychiatric disorders) | 9 (18)
diarrhea (Gastrointestinal disorders) | 8 (10)
alkaline phosphatase increase (Investigations) | 8 (13)
depression (Psychiatric disorders) | 2 (4)
confusion (Psychiatric disorders) | 3 (4)
dehydration (Metabolism and nutrition disorders) | 5 (12)
hypokalemia (Metabolism and nutrition disorders) | 3 (4)
fever (General disorders) | 5 (6)
infection (Infections and infestations) | 7 (11)
weight loss (Metabolism and nutrition disorders) | 5 (5)
sweats (Vascular disorders) | 3 (5)
hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
neutrophil count decreased (Investigations) | 4 (6)
hyponatremia (Metabolism and nutrition disorders) | 7 (7)
thrombosis (Vascular disorders) | 3 (4)
hyperuricemia (Metabolism and nutrition disorders) | 2 (5)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
hypertension (Vascular disorders) | 3 (9)
xerostomia (Gastrointestinal disorders) | 2 (2)
elevated transaminases (Metabolism and nutrition disorders) | 8 (8)
hematuria (Renal and urinary disorders) | 3 (3)
urine retention (Renal and urinary disorders) | 3 (3)
renal failure (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes